CLINICAL TRIAL: NCT04994730
Title: Exenteration: Quality of Life Study and Rehabilitation Rate According to the Reconstruction Technique
Brief Title: Exenteration: Quality of Life Study and Rehabilitation Rate According to the Reconstruction Technique (ETRE)
Acronym: ETRE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Other Study IDs: IC 2020-14
Record Dates: First submitted 2021-08-03; First posted 2021-08-06 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Cancer
Keywords: Exenteration; Surgery; Quality of life
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Quality of life according to the reconstruction technique — For this retrospective analysis, 118 patients could be included, 17 of whom had undergone ante-brachial free flap reconstruction, 16 of whom had undergone this reconstruction within the last 2 years.
  The primary endpoint: Analysis of the quality of life score according to the reconstruction technique (free ante-brachial flap versus others) will be performed by a Wilcoxon-Mann-Whitney test.

SUMMARY:
Prospective monocentric quality of life study. Including all patients who have been exentered at the Institut Curie Paris, from January 2004 to December 2019, proposing to compare the reported quality of life of patients according to the reconstruction technique they have undergone.

The sponsor will evaluate the quality of life of our patients by means of two validated questionnaires, in French, in the context of ENT surgery: the FACT-G and FACT-MBIS questionnaires.

DETAILED DESCRIPTION:
It is now obvious to all surgeons involved in the follow-up of these patients that not all orbital reconstruction techniques are equal.

Thus, through this study, The investigators wish to objectively highlight the gain in quality of life and prosthetic equipment in exentered patients, depending on the reconstruction method used.

This prospective study, including all patients who have been exentered at the Institut Curie Paris, from January 2004 to December 2019, proposes to compare the reported quality of life of patients according to the reconstruction technique patients have undergone.

The investigators will evaluate the quality of life of our patients by means of two validated questionnaires, in French, in the context of ENT surgery: the FACT-G and FACT-MBIS questionnaires. The investigators will submit them, after express telephone agreement, by post to all the patients included in our study.

The aim of such a study will therefore be to provide assistance to both surgeons and patients in the choice of an orbital reconstruction technique, by objectively demonstrating the superiority of one technique over the others in terms of quality of life and prosthetic equipment rate.

The patients included in this study will have to answer two questionnaires, submitted by post. This study therefore falls within the framework of minimal or moderate risk studies.

The patients will be informed by telephone interview about the method of writing the questionnaires and their content.

The investigators will pay particular attention to the quality of life of the patients who have benefited from a free ante-brachial flap reconstruction in comparison with other reconstruction techniques; this will constitute the main criterion of our study.

In addition, the collection of pseudo-anonymised computerised data from all the patient files will give rise to a comparison of post-operative healing times, the rate of prosthetic fitting, and the time taken to fit the prosthesis according to the reconstruction techniques. These three factors, already identified in the literature as indicators of good rehabilitationn , will constitute our secondary judgment criteria.

ELIGIBILITY:
Inclusion Criteria:

All patients, living or lost, exentered at the Institut Curie Paris between January 2014 and December 2019,

Exclusion Criteria:

* Persons under court protection.
* Persons not in a condition to give their consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients, living or lost, exentered at the Institut Curie Paris between January 2014 and December 2019,
Sampling Method: Non-Probability Sample
Enrollment: 118 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2022-05-25 (Estimated); Study Completion 2022-05-25 (Estimated)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy: General (FACT-G) | Baseline
  The FACT-G questionnaire consists of 27 general items, with the patient scoring each item on a scale of 0 to 4. The final score is the sum of all the items.
FACT/McGill Body Image Concern Scale - Head and Neck Cancer Version (FACT-MBIS) | Baseline
  The FACT-MBIS questionnaire consists of 21 items related to self-esteem and social comfort, each item is also scored on a scale of 0 to 4. The final score is the sum of all items.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie BADOIS, MD, Principal Investigator — Institut Curie
Locations (1):
- Institut Curie, Paris, France

IPD SHARING:
Plan to Share IPD: No